CLINICAL TRIAL: NCT06192680
Title: A Multicenter, Single-arm Study of Liposomal Irinotecan and Capecitabine Plus Bevacizumab as Second-line Therapy in Metastatic Colorectal Cancer
Brief Title: Liposomal Irinotecan and Capecitabine Plus Bevacizumab as Second-line Therapy in Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yanqiao Zhang, professor, Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-CRC-K05
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer
Keywords: metastatic disease; liposomal irinotecan; second-line therapy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — irinotecan sucrosofate; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- liposomal irinotecan + capecitabine + bevacizumab (Experimental): liposomal irinotecan 70 mg/m², d1 + capecitabine 1000 mg/m² BID, d1~10 + bevacizumab 5mg/kg, d1.
  q2w
  Interventions: Drug: Liposomal irinotecan; Drug: Capecitabine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Liposomal irinotecan — 70 mg/m² IV
  Other Names: nal-IRI
Drug: Capecitabine — 1000 mg/m² PO BID
  Other Names: Xeloda
Drug: Bevacizumab — 5mg/kg IV
  Other Names: Avastin

SUMMARY:
This multicenter, single-arm trial will explore the efficacy and safety of liposomal irinotecan and capecitabine plus bevacizumab as second-line therapy in metastatic colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) has a poor prognosis and poses a serious threat to human health. irinotecan + fluorouracil ± angiogenesis inhibitors are common treatments for advanced CRC. For patients receiving oxaliplatin-based therapy, irinotecan-based therapy is recommended as second-line therapy. Liposomal irinotecan is a new pharmaceutical form of traditional irinotecan. It adopts a special loading technology to encapsulate traditional irinotecan in liposomes, which can avoid its hydrolysis under physiological conditions, increase the affinity with cancer cells, overcome drug resistance, increase the drug uptake by cancer cells, reduce the drug dose, improve the efficacy and reduce the toxic side effects. The aim of this study is to explore the efficacy and safety of liposomal irinotecan+ capecitabine + bevacizumab as second-line treatment for metastatic CRC.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old.
* Histopathologically and/or cytologically confirmed unresectable metastatic colorectal adenocarcinoma, and patients failed or are intolerant to first-line treatment with oxaliplatin ± VEGF/EGFR.
* At least one measurable lesion (according to RECIST v1.1).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 ~ 1.
* The expected survival time ≥3 months.
* Subject has adequate biological parameters as demonstrated by the following: Absolute neutrophil count (ANC) ≥1.5×10^9/L, Platelet count ≥100×10^9/L, Hemoglobin (Hgb) ≥90 g/L.
* Adequate hepatic function as evidenced by: Total bilirubin ≤1.5 × upper limit of normal (ULN), Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN, ≤5 × ULN if liver metastases are present. Serum albumin ≥3 g/dL.
* Adequate renal function as evidenced by serum creatinine (Cr) ≤1.5 × ULN or creatinine clearance ≥60 mL/min. Proteinuria < 2+ (those with proteinuria ≥2+ at baseline had to demonstrate ≤1 g protein per 24 hours).
* Coagulation function: International normalised ratio (INR) ≤1.5, activated partial thromboplastin time (APTT) ≤1.5 × ULN.
* Left ventricular ejection fraction (LVEF) ≥50%.
* Subjects agree to use contraception and are not pregnant or breastfeeding women.
* Agree and be able to comply with the plan during the study period. Provide written informed consent before entering the study screening.

Exclusion Criteria:

* Any other malignancy within 5 years, with the exception of cured in-situ carcinoma or basal cell carcinoma etc.
* Previous treatment with irinotecan/liposomal irinotecan.
* Patients with the primary lesion located in the left colon and RAS/BRAF wild-type who did not use cetuximab on the first line.
* Known as high microsatellite instability (MSI-H) or mismatch repair deficiency (dMMR).
* Massive pleural effusion or ascites requiring intervention.
* Active, uncontrolled bacterial, viral, or fungal infections that require systemic treatment.
* Active HIV infection.
* Combined with uncontrollable systemic diseases within 6 months before the first administration.
* Presence of severe gastrointestinal disease.
* History of major surgery (such as laparotomy, thoracotomy or intestinal resection) within 28 days before the first administration, or plan to undergo major surgery during the study period.
* Presence of interstitial pneumonia or pulmonary fibrosis.
* History of allergy or hypersensitivity to drug or any of their excipients.
* History of pulmonary hemorrhage/hemoptysis ≥Grade 2 (defined as bright red blood of at least 2.5mL) within one month before the first administration.
* Presence of arterial embolism, severe bleeding (excluding bleeding caused by surgery) or tendency for existing embolism or severe bleeding within 6 months before the first administration.
* Combined symptomatic brain metastasis, meningeal metastasis, spinal cord tumor invasion, and spinal cord compression syndrome.
* Use of strong inhibitors or inducers of CYP3A4, CYP2C8 and UGT1A1 within 14 days before the first administration.
* Use other study drug within 1 month before the first administration.
* Patients who are not suitable to participate in this trial for any reason judged by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression free Survival | 1 year
  Defined as the time between signing the informed consent form to the disease progression (according to RECIST v1.1 criteria) or death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate | 6 months
  Defined as the proportion of patients who achieved complete response (CR) and partial response (PR) according to RECIST v1.1.
Disease Control Rate | 6 months
  Defined as the proportion of patients who achieved complete response (CR), partial response (PR), and stable disease (SD) according to RECIST v1.1.
Duration of Response | 6 months
  Defined as the time from response(when CR or PR is first diagnosed) to disease progression or death due to any cause.
Overall survival | 2 years
  Defined as the time between signing the informed consent form to death due to various causes.
Incidence of adverse events | 7 months
  Use NCI-CTCAE version 5.0 for classification and grading.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqiao Zhang, Professor, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University

IPD SHARING:
Plan to Share IPD: No